CLINICAL TRIAL: NCT03407053
Title: Effect of Ultra Processed Versus Unprocessed Diets on Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 180044; 18-DK-0044 (Other: NIH Clinical Center)
Record Dates: First submitted 2018-01-20; First posted 2018-01-23 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-01-28

CONDITIONS: Healthy Diet
Keywords: Calories; Food Intake; Glucose; Body Composition; Body Weight Regulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-processed diet then unprocessed diet (Active Comparator): Participants assigned to this arm will consume ultra-processed diet for two weeks followed by unprocessed diet for two weeks
  Interventions: Dietary Supplement: Ultra-processed diet; Dietary Supplement: Unprocessed diet
- Unprocessed diet then ultra-processed diet (Active Comparator): Participants assigned to this arm will consume unprocessed diet for two weeks followed by ultra-processed diet for two weeks
  Interventions: Dietary Supplement: Ultra-processed diet; Dietary Supplement: Unprocessed diet

INTERVENTIONS:
Dietary Supplement: Ultra-processed diet — Consuming ultra-processed diet over a 2-week period
Dietary Supplement: Unprocessed diet — Consuming unprocessed diet over a 2-week period

SUMMARY:
Background:

Eating too much processed food is believed to lead to obesity. But the effect of processed food on energy intake has not been carefully studied. Researchers want to study people s diets for 4 weeks and do specialized tests of the effects. Participants will get two diets. They will have the same calories and nutrients, but one diet will be unprocessed food and the other will be ultra-processed.

Objective:

To better understand how processed and unprocessed foods affect daily food consumption and how the body handles blood sugar.

Eligibility:

Healthy adults ages 18-50 who have stable weight and can exercise

Design:

Participants will not eat for 12 hours. Then they will be screened with:

* Medical history
* Physical exam
* Heart and blood tests
* Resting energy expenditure test (REE). A hood will collect air exhaled while lying down for 30-40 minutes.
* Psychiatric questions
* Questions about mood, eating, sleep, and socioeconomic status
* 20-minute stationary biking

Female participants will have a urine pregnancy test.

Participants will stay in the clinic for 4 weeks. For 2 weeks they will get a processed diet. For the other 2 weeks they will get an unprocessed diet. Participants cannot use the study period to gain or lose weight.

Participants will have:

* Meals and snacks provided
* Daily exercise
* Blood, urine, and saliva tests
* To drink a special water and a very sweet liquid
* REE
* Scans and X-rays
* To wear activity monitors and a device to measure blood sugar
* Several 24-hour periods in a room that measures oxygen and carbon dioxide
* Repeats of screening questions
* Questions about hunger and meals
* Sleep monitoring
* Taste tests

DETAILED DESCRIPTION:
Overconsumption of foods that result from extensive industrial processing is believed to contribute to the development of obesity. Ultra-processed foods now represent most of the calories consumed in America and their contribution to overall diet has increased in parallel with the rise in the prevalence of obesity over the past several decades. While such correlations are suggestive, the effect of industrial processing per se, independent of dietary macronutrient composition, on ad libitum energy intake has not been carefully investigated. Therefore, we will conduct feeding studies in adult men and women to investigate the differences in ad libitum energy intake resulting from consuming test diets for a pair of 2-week periods in a randomized, crossover design during a single 4-week period. The test diets presented to participants will be matched for calories, macronutrient composition, sugar, fiber, and sodium, but one diet will be composed of ultra-processed foods whereas the other diet will be unprocessed foods.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults age 18-50 years, male and female
  2. Weight stable (< +/- 5 % over past 6 months)

  4. Body mass index (BMI) greater than or equal to 18 kg/m^2

  5. Willing to cease their habitual caffeine intake during the study, beginning one week prior to inpatient admission

  6. Written informed consent

  7. Willing to eat the food provided in the study

  8. Able to complete daily bouts of stationary cycling at a moderate rate and intensity with a heart rate (HR) equal to or greater than 0.3x(220-age-HR(rest))+HR(rest) but not exceeding 0.4x(220-age-HR(rest))+HR(rest) and no signs of arrhythmia

EXCLUSION CRITERIA:

1. Evidence of metabolic or cardiovascular disease, or disease that may influence metabolism (e.g. cancer, diabetes, thyroid disease)
2. Taking any prescription medication or other drug that may influence metabolism (e.g. diet/weight-loss medication, asthma medication, blood pressure medication, psychiatric medications, corticosteroids, or other medications at the discretion of the PI and/or study team)
3. Hematocrit < 34% (women only)
4. Hematocrit < 40% (men only)
5. Pregnancy, lactation (women only)
6. Participating in a regular exercise program (> 2h/week of vigorous activity)
7. Caffeine consumption > 300 mg/day
8. Regular use of alcohol (> 2 drinks per day), tobacco (smoking or chewing) amphetamines, cocaine, heroin, or marijuana over past 6 months
9. Eating disorders or psychological conditions, such as (but not limited to) claustrophobia, clinical depression, bi-polar disorders, that would be incompatible with safe and successful participation in this study, as determined by investigators.

   --Past or present history of claustrophobia since part of the protocol will involve being confined to a small room for whole-body indirect calorimetry and being in an MRI scanner for liver fat measures
10. Implants, devices, or foreign objects implanted in the body that interfere with the Magnetic Resonance procedures
11. Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, food allergies)
12. Volunteers unwilling or unable to give informed consent
13. Non-English speakers due to unavailability of required questionnaires in other languages.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hall, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Result] Hall KD, Ayuketah A, Brychta R, Cai H, Cassimatis T, Chen KY, Chung ST, Costa E, Courville A, Darcey V, Fletcher LA, Forde CG, Gharib AM, Guo J, Howard R, Joseph PV, McGehee S, Ouwerkerk R, Raisinger K, Rozga I, Stagliano M, Walter M, Walter PJ, Yang S, Zhou M. Ultra-Processed Diets Cause Excess Calorie Intake and Weight Gain: An Inpatient Randomized Controlled Trial of Ad Libitum Food Intake. Cell Metab. 2019 Jul 2;30(1):67-77.e3. doi: 10.1016/j.cmet.2019.05.008. Epub 2019 May 16. PMID 31105044
- [Derived] Brunstrom JM, Schatzker M, Rogers PJ, Courville AB, Hall KD, Flynn AN. Consuming an unprocessed diet reduces energy intake: a post-hoc analysis of an randomized controlled trial reveals a role for human "nutritional intelligence". Am J Clin Nutr. 2025 Dec 29:101183. doi: 10.1016/j.ajcnut.2025.101183. Online ahead of print. PMID 41475551
- [Derived] Abar L, Steele EM, Lee SK, Kahle L, Moore SC, Watts E, O'Connell CP, Matthews CE, Herrick KA, Hall KD, O'Connor LE, Freedman ND, Sinha R, Hong HG, Loftfield E. Identification and validation of poly-metabolite scores for diets high in ultra-processed food: An observational study and post-hoc randomized controlled crossover-feeding trial. PLoS Med. 2025 May 20;22(5):e1004560. doi: 10.1371/journal.pmed.1004560. eCollection 2025 May. PMID 40392756
- [Derived] Hengist A, Ong JA, McNeel K, Guo J, Hall KD. Imprecision nutrition? Intraindividual variability of glucose responses to duplicate presented meals in adults without diabetes. Am J Clin Nutr. 2025 Jan;121(1):74-82. doi: 10.1016/j.ajcnut.2024.10.007. Epub 2024 Dec 2. PMID 39755436
- [Derived] Sciarrillo CM, Guo J, Hengist A, Darcey VL, Hall KD. Diet order significantly affects energy balance for diets varying in macronutrients but not ultraprocessing in crossover studies without a washout period. Am J Clin Nutr. 2024 Oct;120(4):953-963. doi: 10.1016/j.ajcnut.2024.08.013. Epub 2024 Aug 18. PMID 39163976
- [Derived] Sciarrillo CM, Guo J, Hengist A, Darcey VL, Hall KD. Diet order affects energy balance in randomized crossover feeding studies that vary in macronutrients but not ultra-processing. medRxiv [Preprint]. 2023 Oct 4:2023.10.03.23296501. doi: 10.1101/2023.10.03.23296501. PMID 37986904
- [Derived] O'Connor LE, Hall KD, Herrick KA, Reedy J, Chung ST, Stagliano M, Courville AB, Sinha R, Freedman ND, Hong HG, Albert PS, Loftfield E. Metabolomic Profiling of an Ultraprocessed Dietary Pattern in a Domiciled Randomized Controlled Crossover Feeding Trial. J Nutr. 2023 Aug;153(8):2181-2192. doi: 10.1016/j.tjnut.2023.06.003. Epub 2023 Jun 3. PMID 37276937
- [Derived] Jaime-Lara RB, Franks AT, Agarwal K, Nawal N, Courville AB, Guo J, Yang S, Brooks BE, Roy A, Taylor K, Darcey VL, LeCheminant JD, Chung S, Forde CG, Hall KD, Joseph PV. No significant salt or sweet taste preference or sensitivity differences following ad libitum consumption of ultra-processed and unprocessed diets: a randomized controlled pilot study. Chem Senses. 2023 Jan 1;48:bjad007. doi: 10.1093/chemse/bjad007. PMID 36897799
- [Derived] Howard R, Guo J, Hall KD. Imprecision nutrition? Different simultaneous continuous glucose monitors provide discordant meal rankings for incremental postprandial glucose in subjects without diabetes. Am J Clin Nutr. 2020 Oct 1;112(4):1114-1119. doi: 10.1093/ajcn/nqaa198. PMID 32766882
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-DK-0044.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultra-processed Diet Then Unprocessed Diet | Unprocessed Diet Then Ultra-processed Diet
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultra-processed Diet Then Unprocessed Diet | Unprocessed Diet Then Ultra-processed Diet | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (6.8) | 30.1 (7.8) | 31.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 2 | 1 | 3
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Body weight [Mean (Standard Deviation); unit: kg] — Body weight in kg
  kg | 77.3 (21.1) | 79.3 (22.4) | 78.3 (21.2)
Fat mass [Mean (Standard Deviation); unit: kg] — Fat mass measured in kilograms (kg). Body fat mass was measured using Dual-energy X-ray absorptiometry (DXA) measurements.
  kg | 23.1 (13.4) | 26.0 (14.2) | 24.6 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: Ad Libitum Energy Intake
Description: Ad libitum energy intake averaged over 14 days for each diet, measured in kilocalories (kcal) per day.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: kcal per day
Groups:
- Ultra-processed Diet: Consuming ultra-processed diet over a 14 day period
- Unprocessed Diet: Consuming unprocessed diet over a 14 day period
Arm/Group | Ultra-processed Diet | Unprocessed Diet
Number analyzed (Participants) | 20 | 20
kcal per day | 2963 (74.3) | 2491 (74.3)

2. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to day 14 for each diet, measured in kilograms (kg)
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: kg
Arm/Group | Ultra-processed Diet | Unprocessed Diet
Number analyzed (Participants) | 20 | 20
kg | 0.94 (0.31) | -0.91 (0.31)

3. Secondary Outcome: Change in Fat Mass
Description: Change in body fat mass from baseline to day 14 for each diet, measured in kilograms (kg). Body fat mass was measured using Dual-energy X-ray absorptiometry (DXA) measurements.
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: kg
Arm/Group | Ultra-processed Diet | Unprocessed Diet
Number analyzed (Participants) | 20 | 19
kg | 0.43 (0.11) | -0.28 (0.11)

ADVERSE EVENTS:
Time Frame: During each 14 day diet period
Arm/Group | Ultra-processed Diet | Unprocessed Diet
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT03407053/Prot_SAP_000.pdf